CLINICAL TRIAL: NCT03527173
Title: Efficacy, Safety and Immunogenicity of GVGH Shigella Sonnei Vaccine (1790GAHB) in a Human Challenge Study of Healthy Non-immune Adults
Brief Title: A Study to Evaluate the Efficacy, Safety and Immunogenicity of a Vaccine Designed to Protect Against Infection With Shigella Sonnei in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205626; H03_03TP (Other: GSK Vaccines Institute for Global Health)
Record Dates: First submitted 2018-05-04; First posted 2018-05-17 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Dysentery, Bacillary
Keywords: Challenge; Efficacy; Shigellosis; Vaccination
MeSH Terms: conditions — Dysentery, Bacillary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind The subject, the site and sponsor personnel involved in the clinical evaluation of the subjects are blinded while other study personnel may be aware of the treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- S. sonnei Group (Experimental): Male or female subjects between, and including, 18 and 50 years of age at the time of the first vaccination, received 2 doses of the S. sonnei study vaccine at Day 1 and Day 29 respectively, by intramuscular injection into the upper deltoid region of the non-dominant arm. At 28 days after the second dose (Day 57), subjects received the challenge dose of S. sonnei 53G strain, orally.
  Interventions: Biological: S.sonnei vaccine; Biological: S. sonnei 53G challenge strain
- Placebo Group (Placebo Comparator): Male or female subjects between, and including, 18 and 50 years of age at the time of the first vaccination, received 2 doses of the placebo at Day 1 and Day 29 respectively, by intramuscular injection into the upper deltoid region of the non-dominant arm. At 28 days after the second dose (Day 57), subjects received the challenge dose of S. sonnei 53G strain, orally.
  Interventions: Drug: Placebo; Biological: S. sonnei 53G challenge strain

INTERVENTIONS:
Biological: S.sonnei vaccine — Subjects receiving 2 doses of the study vaccine by intramuscular route, 28 days apart (at Day 1 and Day 29).
  Other Names: GSK3536852A vaccine
  Arms: S. sonnei Group
Drug: Placebo — Subjects receiving 2 doses of placebo by intramuscular route, 28 days apart (at Day 1 and Day 29).
  Other Names: GAHB-Placebo
  Arms: Placebo Group
Biological: S. sonnei 53G challenge strain — Subjects receiving the challenge dose of S. sonnei 53G strain, orally, at Day 57.

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety and immunogenicity of the GSK3536852A vaccine, which was designed to protect against shigellosis caused by Shigella sonnei (S. sonnei) and is using the new Generalized Modules for Membrane Antigens (GMMA) platform technology developed by GlaxoSmithKline (GSK) Vaccines Institute for Global Health (GVGH).

The study vaccine could be the stepping stone for the development of a multivalent broadly protective Shigella vaccine for vaccination of impoverished communities where shigellosis is endemic. However, a standalone monovalent vaccine against S. sonnei could be used to protect travelers against diarrheal shigellosis, as the vast majority of travelers' shigellosis is caused by S. sonnei, and even to protect infants in endemic regions where shigellosis is primarily caused by S. sonnei.

The GSK3536852A vaccine has been tested in two Phase I dose escalation studies in Europe to assess its safety and immunogenicity via three routes of administration: intramuscular (IM), intranasal (IN) and intradermal (ID). The results from the first study (dose escalation with IM vaccination) have shown that the vaccine has an acceptable safety profile and is well-tolerated up to a dose of 100 micrograms (µg). The results from the second study (dose escalation with ID, IN and IM vaccination) showed that GSK3536852A vaccine is well-tolerated also when administered by the ID and IN routes of vaccination. However, immunogenicity data have shown that GSK3536852A vaccine administered by the ID and IN routes is not as immunogenic as GSK3536852A vaccine administered by the IM route. Therefore, it has been decided to proceed with the clinical development program of this vaccine only using the IM vaccination route. In terms of dosage, the regimen tested in Phase I studies (three doses given one month apart) did not show any significant benefit from the third dose in terms of immunogenicity, therefore a two dose schedule was selected for next studies.

A Phase IIa study, conducted in endemic regions of Africa (i.e., Kenya), has been completed and confirmed the acceptable safety profile and immunogenicity of GSK3536852A vaccine.

Performing this vaccine-human challenge study may give the opportunity to establish evidence of clinical protection induced by the candidate S. sonnei vaccine (GSK3536852A vaccine) at an early development stage.

DETAILED DESCRIPTION:
The original study protocol has been amended due to requests from the Food and Drug Administration (FDA), requests from the funder of the study, Bill & Melinda Gates Foundation (BMGF), to add an additional interim analysis for immunogenicity data that will accelerate the release of key results to help the planning of other studies, and to further align the protocol to other GSK studies and to the challenge model established at the Cincinnati Children's Hospital Medical Centre.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* Individuals who, after the nature of the study has been explained to them, have shown adequate comprehension of the study procedures and knowledge of study.
* A male or female between, and including, 18 and 50 years of age at the time of the first vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Seronegative for human immunodeficiency virus (HIV), hepatitis B and C.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * Has practiced adequate contraception for 30 days prior to vaccination, and
  * Has a negative pregnancy test on the day of vaccination, and
  * Has agreed to continue adequate contraception during the entire study period.

Exclusion Criteria:

* Received an investigational or non-registered medicinal product within 30 days prior to informed consent, or planned use during the study period.
* Any behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
* History of any neurological disorders or seizures.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the subject due to participation in the study.
* Human Leukocyte Antigen (HLA)-B27 positive test at screening and/or with history of reactive arthritis.
* Clinical conditions representing a contraindication to intramuscular vaccination and blood draws.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine/placebo dose. For corticosteroids, this will mean prednisone ≥ 20 milligrams (mg)/day, or equivalent. Inhaled except for doses > 800 µg/day and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period. Subjects may be on chronic or as needed medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition.
* Known bleeding diathesis or any condition that may be associated with a prolonged bleeding time.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* History of having participated in a previous Shigella challenge study.
* Individuals who have a previously laboratory confirmed case of disease caused by S. sonnei or serology positive for local anti S. sonnei LPS IgG Screening-ELISA at screening.
* History of any serious chronic or progressive disease according to judgment of the investigator.
* History of any malignancy or lymphoproliferative disorder.
* Known to be part of study personnel or being a close family member to the personnel conducting this study.
* History of anaphylactic reaction or allergy to vaccine/placebo or challenge agent components or any other allergies deemed by the investigator to increase the risk of an AE if they were to participate in the study.
* Known allergy to ciprofloxacin or the other antibiotics used for treatment as deemed by the investigator.
* Individuals receiving a course of antibiotics within a week of the challenge will be ineligible to receive the challenge strain.
* History of gastric acid hyper-secretory disorders as assessed and judged by the investigator or any other significant intestinal disorder.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine/placebo or challenge agent.
* Acute disease and/or fever at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests. Chronic medical diagnoses or conditions should be stable for the last 60 days. This includes no change in chronic prescription medication, dose, or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrolment.
* A clinically significant sign or symptoms of acute illness, significant anomalies in vital signs.
* Known to handle food as part of work related activities.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Received immunoglobulins or any blood products within 180 days prior to informed consent or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* Females with history of stillbirth, neonatal loss, or previous infant with anomaly, except those who have had a planned termination of pregnancy, hysterectomy or bilateral tubal ligation.
* History of chronic alcohol consumption and/or drug abuse. Chronic alcohol consumption is defined as: a prolonged period of frequent, heavy alcohol use; the inability to control drinking once it has begun; physical dependence manifested by withdrawal symptoms when the individual stops using alcohol; tolerance, or the need to use more and more alcohol to achieve the same effects; a variety of social and/or legal problems arising from alcohol use.
* Known to have close household or professional contacts with people with immunosuppressive condition.
* Documented HIV, hepatitis B and C positive subject.
* Any condition which, in the opinion of the investigator, may pose an increased and unreasonable safety risk to the subject if they participated in the study.
* Subjects with a baseline neutrophil count below 1800 cells per microliter (cells/µL) lower limit of normal range (LLN) OR with clinically significant abnormalities in other laboratory values, according to local reference ranges and investigator judgment.
* Previous history of Benign Ethnic Neutropenia, or drug related Neutropenia.
* Concomitant treatment with neutropenic agents.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-05-08 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at one center in the United States of America (USA).
Pre-assignment Details: All 71 subjects enrolled in the study, received a study vaccination and were included in the All Exposed Set.
Period: Overall Study
Arm/Group | S. Sonnei Group | Placebo Group
Started | 36 | 35
Completed | 29 | 28
Not Completed | 7 | 7
Not completed — Lost to Follow-up | 4 | 2
Not completed — ELIGIBILITY CRITERIA NOT FULFILLED | 1 | 0
Not completed — CONSENT WITHDRAWAL NOT DUE TO ADV. EVENT | 1 | 5
Not completed — NOT WILLING TO PARTICIPATE THIS VISIT | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | S. Sonnei Group | Placebo Group | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.2 (9.9) | 35.2 (8.5) | 35.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 22 | 18 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 24 | 28 | 52
  OTHER - UNSPECIFIED | 2 | 1 | 3
  WHITE | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With at Least One Episode of Shigellosis According to the Protocol Primary Case Definition
Description: Attack rate of shigellosis expressed as percentage of subjects with at least one episode of shigellosis after challenge, and 90% confidence interval (CI) (Clopper-Pearson method). Episodes of shigellosis fulfilling primary case definition: Shedding of S. sonnei 53G accompanied by moderate or severe diarrhea OR shedding with oral temperature greater than or equal to (≥) 38.5°C. Moderate diarrhea consists of 4 to 5 loose or watery (Grade [G]3 to 5) stools or 400 to 800 grams of G3 to 5 stools within 24 hours. Severe diarrhea consists of 6 or more loose or watery (G3 to 5) stools or > 800 grams of G3 to 5 stools within 24 hours or required medical intervention. In case of severe diarrhea, medical intervention is defined as intravenous fluids administration or anticipation of antibiotic treatment before the 5th day after challenge. G3 = viscous opaque liquid or semi-liquid which assumes the shape of the bowl; G4 = watery opaque liquid; G5 = clear watery or mucoid liquid.
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: The analysis is performed on the Per-protocol set (PPS) for efficacy, which includes all subjects who received the study vaccine or placebo according to protocol, were not excluded due to other reasons defined prior to unblinding or analysis and who received the challenge agent.
Measure: Number (90% Confidence Interval); unit: Percentage of subjects
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 32 | 28
Percentage of subjects | 46.9 [31.5 to 62.7] | 42.9 [26.9 to 60.0]
Statistical Analysis 1: Comparison: S. Sonnei Group vs Placebo Group; To demonstrate the efficacy of two vaccinations with 25 µg of S. sonnei vaccine in healthy adults compared to placebo in preventing shigellosis, fulfilling the protocol primary case definition, after challenge with S. sonnei 53G strain. Vaccine efficacy (VE) rate was assessed as 1-Risk Ratio(RR) with RR = ratio of proportion of subjects with shigellosis in the vaccinated group on the proportion of subjects with shigellosis in the placebo group; Test type: Non-Inferiority — VE in reduction of shigellosis is demonstrated if lower limit (LL) of 90% CI of VE estimated with Miettinen-Nurminen (M-N) method is above 0. This estimated CI was complemented with Barnard test. The LL of the 90% CI for VE calculated with M-N method is above 0 if the p-value of the one-sided Barnard test is below 5%; p = 0.4266, 1-sided Barnard Unconditional Exact Test; Vaccine efficacy rate = -9.4, 90% CI 2-sided [-96.7 to 33.7]

2. Secondary Outcome: Percentage of Subjects With at Least One Episode of Shigellosis According to Controlled Human Infection Model (CHIM) Working Group Case Definition for Shigellosis
Description: Percentage of subjects with shigellosis fulfilling the CHIM expert working group case definition for shigellosis, and 90% confidence interval (CI) (Clopper-Pearson method). According to the working group, the participant must fulfil any of the three following possible endpoints to qualify as having reached the CHIM case definition for this objective: 1. Severe diarrhea defined as [[≥ 6 loose stools in 24 hours] OR [˃800 grams loose stools in 24 hours]; 2. Moderate diarrhea defined as [4-5 loose stools in 24 hours OR 400-800 grams loose stools in 24 hours] AND [oral temperature [≥ 38.0°C OR [≥ 1 moderate constitutional/enteric symptom OR [≥ 2 episodes of vomiting in 24 hours]; 3. Dysentery defined as [[≥ 2 loose stools with gross blood (hemoccult positive) in 24 hours] AND [oral temperature [≥ 38.0°C OR [≥ 1 moderate constitutional/enteric symptom OR [≥ 2 episodes of vomiting in 24 hours].
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of subjects
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 32 | 28
Percentage of subjects | 46.9 [31.5 to 62.7] | 32.1 [17.9 to 49.4]

3. Secondary Outcome: Percentage of Subjects With at Least One Episode of Shigellosis
Description: Percentage of subjects with shigellosis fulfilling the following definition of shigellosis (with 90% confidence interval (CI) - Clopper-Pearson method): 1) severe diarrhea OR 2) moderate diarrhea AND oral temperature ≥ 38.0 °C OR ≥ 1 moderate constitutional/enteric symptom OR 3) dysentery [[≥ 2 loose stools with gross blood (hemoccult positive) in 24 hours] AND [≥ 1 reportable constitutional/enteric symptom]].
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of subjects
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 32 | 28
Percentage of subjects | 46.9 [31.5 to 62.7] | 35.7 [20.8 to 53.0]

4. Secondary Outcome: Percentage of Subjects With at Least One Episode of More Severe Shigellosis
Description: Percentage of subjects with more severe shigellosis fulfilling the following definition of more severe shigellosis (with 90% confidence interval (CI) - Clopper-Pearson method): 1) moderate OR severe diarrhea AND oral temperature ≥ 38.0 °C OR ≥ 1 severe constitutional/enteric symptom OR 2) dysentery [[≥ 2 loose stools with gross blood (hemoccult positive) in 24 hours] AND [oral temperature ≥ 38.0°C OR ≥ 1 severe constitutional/enteric symptom]].
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of subjects
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 32 | 28
Percentage of subjects | 15.6 [6.4 to 30.1] | 14.3 [5.0 to 29.8]

5. Secondary Outcome: Percentage of Subjects With Specific Disease Symptoms
Description: Percentage of subjects with 90% CI-Clopper-Pearson method was also measured for: shedding of S.sonnei strain 53G (defined as positivity of ≥1 stool sample by culture/quantitative Polymerase Chain Reaction/both); severe diarrhea; more severe diarrhea; dysentery; confirmed S.sonnei 53G shedding AND moderate or severe diarrhea OR dysentery OR presence of oral temperature ≥ 38.5°C OR presence of 1 or more severe intestinal symptoms (abdominal pain, cramping, nausea, vomiting, gas, and anorexia) abbreviated as "shedding of S.sonnei 53G and […"; disease not fulfilling the protocol primary case definition for shigellosis associated or not with mild to moderate symptoms including: ≥1 stool and no moderate or severe diarrhea evidence, abdominal pain, abdominal cramps, gas, anorexia, nausea, headache, myalgia, malaise, arthralgia, fever, vomiting and intravenous fluid administration. Any=any symptom regardless of intensity grade or relation to study vaccination and/or challenge administration.
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percentage of subjects
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 32 | 28
Percentage of subjects
  Shedding of S. sonnei strain 53G | 96.9 [86.0 to 99.8] | 100 [89.9 to 100.0]
  Severe diarrhea | 40.6 [26.0 to 56.7] | 25 [12.4 to 41.9]
  More severe diarrhea | 34.4 [20.6 to 50.4] | 17.9 [7.3 to 33.9]
  Dysentery | 34.4 [20.6 to 50.4] | 28.6 [15.1 to 45.7]
  Shedding of S. sonnei 53G and [… | 46.9 [31.5 to 62.7] | 42.9 [26.9 to 60.0]
  ≥1 stool and no moderate/severe diarrhea evidence | 50.0 [34.4 to 65.6] | 60.7 [43.5 to 76.2]
  Any Abdominal pain | 50.0 [34.4 to 65.6] | 46.4 [30.1 to 63.4]
  Any Abdominal cramps | 53.1 [37.3 to 68.5] | 50.0 [33.3 to 66.7]
  Any Gas | 40.6 [26.0 to 56.7] | 57.1 [40.0 to 73.1]
  Any Anorexia | 43.8 [28.7 to 59.7] | 46.4 [30.1 to 63.4]
  Any Nausea | 34.4 [20.6 to 50.4] | 32.1 [17.9 to 49.4]
  Any Headache | 53.1 [37.3 to 68.5] | 60.7 [43.5 to 76.2]
  Any Myalgia | 34.4 [20.6 to 50.4] | 46.4 [30.1 to 63.4]
  Any Malaise | 46.9 [31.5 to 62.7] | 57.1 [40.0 to 73.1]
  Any Arthralgia | 28.1 [15.5 to 43.9] | 32.1 [17.9 to 49.4]
  Any Fever | 9.4 [2.6 to 22.5] | 17.9 [7.3 to 33.9]
  Any Vomiting | 21.9 [10.7 to 37.2] | 7.1 [1.3 to 20.8]
  Intravenous fluid administration | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]

6. Secondary Outcome: Mean Number of Grade 3-5 Stools Per Subject
Description: The mean number of grade 3-5 stools (and standard deviation) were calculated per subject from challenge to discharge.
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grade 3-5 stools
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 32 | 28
grade 3-5 stools | 28 (13.0) | 13.9 (6.6)

7. Secondary Outcome: Weight of Grade 3-5 Stools
Description: Mean and standard deviation (SD) of weights were expressed in grams. The following measures were calculated: mean and SD of the weight of grade 3-5 stools calculated on all subjects (Weight/all subjects), mean and SD of the weight of grade 3-5 stools calculated on subjects with at least one grade 3-5 stool (Weight/subj.with at least 1 grade 3-5 stool), Cumulative mean and SD weight of grade 3-5 stools per subjects, accumulated from challenge to discharge (Cumulative weight/all subjects).
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Grams
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 32 | 28
Grams
  Weight/all subjects | 87.4 (68.3) | 91.3 (54.7)
  Weight/subj. with at least 1 grade 3-5 stool: number analyzed (Participants) | 22 | 22
  Weight/subj. with at least 1 grade 3-5 stool | 127.2 (39.8) | 116.3 (28.5)
  Cumulative weight/all subjects | 1161.1 (1416.9) | 766.9 (884.9)

8. Secondary Outcome: Time (Days) From Challenge Administration to Onset of Shigellosis, According to the Primary Case Definition
Description: Median time to onset of shigellosis was to be estimated with Kaplan-Meier method among subjects who received the challenge agent. The day associated to the first shigellosis was the time of onset of shigellosis. Subjects who did not have shigellosis were censored at the time on the day of discharge. Median time (in days) to onset of shigellosis and 90% confidence interval (CI) could not be calculated in any of the groups because less than 50% of subjects experienced the event (shigellosis) during the observation period.
Time Frame: Starting with the challenge visit (Day 57) and lasting up to the end of the inpatient stay (Day 64)
Population: The analysis was not performed because less than 50% of subjects experienced the event (shigellosis) during the observation period. Therefore, the Median time to onset of shigellosis and 90% confidence interval (CI) could not be calculated in any of the groups.
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs)
Description: Solicited local AEs include: pain, erythema and induration at injection site. Any = occurrence of local adverse event regardless of intensity grade. Any erythema or induration at injection site is any symptom with a surface diameter greater than 25 millimeters.
Time Frame: During the 7-day period after each vaccination (vaccine/placebo administered at Day 1 and Day 29)
Population: The analysis is performed on Solicited Safety Set, which includes all enrolled subjects who received the study vaccine or placebo, with valid data on solicited AEs and with the Subject Diary completed.
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 36 | 35
Participants
  Dose 1, Pain | 29 | 12
  Dose 2, Pain: number analyzed (Participants) | 36 | 34
  Dose 2, Pain | 24 | 5
  Dose 1, Erythema | 0 | 0
  Dose 2, Erythema: number analyzed (Participants) | 36 | 34
  Dose 2, Erythema | 0 | 0
  Dose 1, Induration | 0 | 1
  Dose 2, Induration: number analyzed (Participants) | 36 | 34
  Dose 2, Induration | 0 | 0

10. Secondary Outcome: Number of Subjects With Any Solicited Systemic AEs
Description: Solicited systemic AEs include: arthralgia, chills, fatigue, headache, malaise, myalgia, fever (oral temperature ≥ 38.0°C). Any = occurrence of systemic adverse event regardless of intensity and relation to study vaccination.
Time Frame: During the 7-day period after each vaccination (vaccine/placebo administered at Day 1 and Day 29)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 36 | 35
Participants
  Dose 1, Arthralgia | 6 | 3
  Dose 2, Arthralgia: number analyzed (Participants) | 36 | 34
  Dose 2, Arthralgia | 7 | 2
  Dose 1, Chills | 5 | 2
  Dose 2, Chills: number analyzed (Participants) | 36 | 34
  Dose 2, Chills | 3 | 1
  Dose 1, Fatigue | 6 | 8
  Dose 2, Fatigue: number analyzed (Participants) | 36 | 34
  Dose 2, Fatigue | 7 | 3
  Dose 1, Headache | 10 | 8
  Dose 2, Headache: number analyzed (Participants) | 36 | 34
  Dose 2, Headache | 4 | 4
  Dose 1, Malaise | 8 | 4
  Dose 2, Malaise: number analyzed (Participants) | 36 | 34
  Dose 2, Malaise | 6 | 4
  Dose 1, Myalgia | 15 | 8
  Dose 2, Myalgia: number analyzed (Participants) | 36 | 34
  Dose 2, Myalgia | 9 | 7
  Dose 1, Fever | 1 | 0
  Dose 2, Fever: number analyzed (Participants) | 36 | 34
  Dose 2, Fever | 0 | 0

11. Secondary Outcome: Number of Subjects With Any Unsolicited AEs During the 28-day Post-vaccination Period
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to study vaccination.
Time Frame: During the 28-day period across doses (vaccine/placebo administered at Day 1 and Day 29)
Population: The analysis is performed on the Unsolicited Safety Set, which includes all enrolled subjects who received the study vaccine or placebo, with unsolicited AE data.
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 36 | 34
Participants | 18 | 13

12. Secondary Outcome: Number of Subjects With Any Unsolicited AEs During the 28-day Follow-up Period After Challenge
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to study vaccination and/or challenge agent administration.
Time Frame: During the 28-day follow-up period after challenge (challenge administered at Day 57)
Population: The analysis is performed on the Unsolicited Safety Set, which includes all enrolled subjects who received the study vaccine or placebo, and the challenge agent administration, and with unsolicited AE data.
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 33 | 29
Participants | 20 | 17

13. Secondary Outcome: Number of Subjects With Any Serious Adverse Events (SAEs) and Related SAEs
Description: Serious adverse events (SAEs) assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity. Related SAEs = SAEs assessed by the investigator as related to the study vaccination and/or challenge agent administration.
Time Frame: From Day 1 up to study end at Day 237
Population: The analysis is performed on the Overall Safety Set, which includes all enrolled subjects who received the study vaccine or placebo, and who are in the Solicited Safety Set and/or Unsolicited Safety Set.
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 36 | 35
Participants
  Any SAE(s) | 0 | 1
  Related SAE(s) | 0 | 0

14. Secondary Outcome: Number of Subjects With Any Adverse Events of Special Interest (AESI) (i.e., Symptomatic Neutropenia)
Description: AESI are predefined (serious or non-serious) AEs of scientific and medical concern specific to the product or program, for which ongoing monitoring and rapid communication by the investigator to the sponsor can be appropriate, because such an event might warrant further investigation in order to characterize and understand it.
Time Frame: From Day 1 up to study end at Day 237
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 36 | 35
Participants | 0 | 0

15. Secondary Outcome: Number of Subjects With Change From Baseline in Hematological Laboratory Parameters With Respect to Normal Laboratory Ranges
Description: Among hematological parameters assessed are: Basophils, Eosinophils, Erythrocytes, Hematocrit, Hemoglobin, Leukocytes, Lymphocytes, Monocytes, Neutrophils and Platelets. Below = below the normal laboratory range defined for the specified laboratory parameter; Above = above the normal laboratory range defined for the specified laboratory parameter; Within = within the normal laboratory range defined for the specified laboratory parameter. Category naming has been defined as follows: Parameter, time point, range indicator at Baseline, range indicator at the specified time point: e.g.: "Basophils, Day 8, Within, Within ". Note: All subjects whose neutrophil value was below the threshold defined in the Protocol, at any time during the study, were re-tested until neutropenia resolution.
Time Frame: At Day 8, at Day 36 and at Day 237
Population: The analysis is performed on the Exposed Set, which includes all enrolled subjects who received the study vaccination and with laboratory data for the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 36 | 35
Participants
  Basophils, Day 8, Within, Within: number analyzed (Participants) | 33 | 30
  Basophils, Day 8, Within, Within | 31 | 28
  Basophils, Day 8, Within, Above: number analyzed (Participants) | 33 | 30
  Basophils, Day 8, Within, Above | 2 | 2
  Basophils, Day 8, Above, Within: number analyzed (Participants) | 3 | 5
  Basophils, Day 8, Above, Within | 2 | 5
  Basophils, Day 8, Above, Above: number analyzed (Participants) | 3 | 5
  Basophils, Day 8, Above, Above | 1 | 0
  Basophils, Day 36, Within, Within: number analyzed (Participants) | 33 | 29
  Basophils, Day 36, Within, Within | 32 | 26
  Basophils, Day 36, Within, Above: number analyzed (Participants) | 33 | 29
  Basophils, Day 36, Within, Above | 1 | 3
  Basophils, Day 36, Above, Within: number analyzed (Participants) | 3 | 5
  Basophils, Day 36, Above, Within | 2 | 4
  Basophils, Day 36, Above, Above: number analyzed (Participants) | 3 | 5
  Basophils, Day 36, Above, Above | 1 | 1
  Basophils, Day 237, Within, Within: number analyzed (Participants) | 26 | 24
  Basophils, Day 237, Within, Within | 25 | 22
  Basophils, Day 237, Within, Above: number analyzed (Participants) | 26 | 24
  Basophils, Day 237, Within, Above | 1 | 2
  Basophils, Day 237, Above, Within: number analyzed (Participants) | 3 | 4
  Basophils, Day 237, Above, Within | 3 | 4
  Eosinophils, Day 8, Within, Within: number analyzed (Participants) | 36 | 34
  Eosinophils, Day 8, Within, Within | 35 | 34
  Eosinophils, Day 8, Within, Above: number analyzed (Participants) | 36 | 34
  Eosinophils, Day 8, Within, Above | 1 | 0
  Eosinophils, Day 8, Above, Within: number analyzed (Participants) | 0 | 1
  Eosinophils, Day 8, Above, Within |  | 1
  Eosinophils, Day 36, Within, Within: number analyzed (Participants) | 36 | 33
  Eosinophils, Day 36, Within, Within | 36 | 32
  Eosinophils, Day 36, Within, Above: number analyzed (Participants) | 36 | 33
  Eosinophils, Day 36, Within, Above | 0 | 1
  Eosinophils, Day 36, Above, Within: number analyzed (Participants) | 0 | 1
  Eosinophils, Day 36, Above, Within |  | 1
  Eosinophils, Day 237, Within, Within: number analyzed (Participants) | 29 | 27
  Eosinophils, Day 237, Within, Within | 29 | 27
  Eosinophils, Day 237, Above, Within: number analyzed (Participants) | 0 | 1
  Eosinophils, Day 237, Above, Within |  | 1
  Erythrocytes, Day 8, Below, Below: number analyzed (Participants) | 5 | 0
  Erythrocytes, Day 8, Below, Below | 4 |
  Erythrocytes, Day 8, Below, Within: number analyzed (Participants) | 5 | 0
  Erythrocytes, Day 8, Below, Within | 1 |
  Erythrocytes, Day 8, Within, Below: number analyzed (Participants) | 31 | 33
  Erythrocytes, Day 8, Within, Below | 2 | 2
  Erythrocytes, Day 8, Within, Within: number analyzed (Participants) | 31 | 33
  Erythrocytes, Day 8, Within, Within | 29 | 31
  Erythrocytes, Day 8, Above, Within: number analyzed (Participants) | 0 | 2
  Erythrocytes, Day 8, Above, Within |  | 2
  Erythrocytes, Day 36, Below, Below: number analyzed (Participants) | 5 | 0
  Erythrocytes, Day 36, Below, Below | 4 |
  Erythrocytes, Day 36, Below, Within: number analyzed (Participants) | 5 | 0
  Erythrocytes, Day 36, Below, Within | 1 |
  Erythrocytes, Day 36, Within, Below: number analyzed (Participants) | 31 | 32
  Erythrocytes, Day 36, Within, Below | 2 | 2
  Erythrocytes, Day 36, Within, Within: number analyzed (Participants) | 31 | 32
  Erythrocytes, Day 36, Within, Within | 29 | 30
  Erythrocytes, Day 36, Above, Within: number analyzed (Participants) | 0 | 2
  Erythrocytes, Day 36, Above, Within |  | 2
  Erythrocytes, Day 237, Below, Below: number analyzed (Participants) | 5 | 0
  Erythrocytes, Day 237, Below, Below | 3 |
  Erythrocytes, Day 237, Below, Within: number analyzed (Participants) | 5 | 0
  Erythrocytes, Day 237, Below, Within | 2 |
  Erythrocytes, Day 237, Within, Below: number analyzed (Participants) | 24 | 26
  Erythrocytes, Day 237, Within, Below | 1 | 0
  Erythrocytes, Day 237, Within, Within: number analyzed (Participants) | 24 | 26
  Erythrocytes, Day 237, Within, Within | 22 | 25
  Erythrocytes, Day 237, Within, Above: number analyzed (Participants) | 24 | 26
  Erythrocytes, Day 237, Within, Above | 1 | 1
  Erythrocytes, Day 237, Above, Within: number analyzed (Participants) | 0 | 2
  Erythrocytes, Day 237, Above, Within |  | 1
  Erythrocytes, Day 237, Above, Above: number analyzed (Participants) | 0 | 2
  Erythrocytes, Day 237, Above, Above |  | 1
  Hematocrit, Day 8, Below, Below: number analyzed (Participants) | 4 | 1
  Hematocrit, Day 8, Below, Below | 3 | 1
  Hematocrit, Day 8, Below, Within: number analyzed (Participants) | 4 | 1
  Hematocrit, Day 8, Below, Within | 1 | 0
  Hematocrit, Day 8, Within, Below: number analyzed (Participants) | 32 | 32
  Hematocrit, Day 8, Within, Below | 3 | 1
  Hematocrit, Day 8, Within, Within: number analyzed (Participants) | 32 | 32
  Hematocrit, Day 8, Within, Within | 29 | 31
  Hematocrit, Day 8, Above, Within: number analyzed (Participants) | 0 | 2
  Hematocrit, Day 8, Above, Within |  | 2
  Hematocrit, Day 36, Below, Below: number analyzed (Participants) | 4 | 1
  Hematocrit, Day 36, Below, Below | 2 | 1
  Hematocrit, Day 36, Below, Within: number analyzed (Participants) | 4 | 1
  Hematocrit, Day 36, Below, Within | 2 | 0
  Hematocrit, Day 36, Within, Below: number analyzed (Participants) | 32 | 31
  Hematocrit, Day 36, Within, Below | 3 | 2
  Hematocrit, Day 36, Within, Within: number analyzed (Participants) | 32 | 31
  Hematocrit, Day 36, Within, Within | 29 | 29
  Hematocrit, Day 36, Above, Within: number analyzed (Participants) | 0 | 2
  Hematocrit, Day 36, Above, Within |  | 2
  Hematocrit, Day 237, Below, Below: number analyzed (Participants) | 4 | 0
  Hematocrit, Day 237, Below, Below | 3 |
  Hematocrit, Day 237, Below, Within: number analyzed (Participants) | 4 | 0
  Hematocrit, Day 237, Below, Within | 1 |
  Hematocrit, Day 237, Within, Below: number analyzed (Participants) | 25 | 26
  Hematocrit, Day 237, Within, Below | 1 | 2
  Hematocrit, Day 237, Within, Within: number analyzed (Participants) | 25 | 26
  Hematocrit, Day 237, Within, Within | 24 | 24
  Hematocrit, Day 237, Above, Within: number analyzed (Participants) | 0 | 2
  Hematocrit, Day 237, Above, Within |  | 1
  Hematocrit, Day 237, Above, Above: number analyzed (Participants) | 0 | 2
  Hematocrit, Day 237, Above, Above |  | 1
  Hemoglobin, Day 8, Below, Below: number analyzed (Participants) | 4 | 1
  Hemoglobin, Day 8, Below, Below | 4 | 1
  Hemoglobin, Day 8, Within, Below: number analyzed (Participants) | 32 | 34
  Hemoglobin, Day 8, Within, Below | 3 | 2
  Hemoglobin, Day 8, Within, Within: number analyzed (Participants) | 32 | 34
  Hemoglobin, Day 8, Within, Within | 29 | 32
  Hemoglobin, Day 36, Below, Below: number analyzed (Participants) | 4 | 1
  Hemoglobin, Day 36, Below, Below | 3 | 1
  Hemoglobin, Day 36, Below, Within: number analyzed (Participants) | 4 | 1
  Hemoglobin, Day 36, Below, Within | 1 | 0
  Hemoglobin, Day 36, Within, Below: number analyzed (Participants) | 32 | 33
  Hemoglobin, Day 36, Within, Below | 3 | 1
  Hemoglobin, Day 36, Within, Within: number analyzed (Participants) | 32 | 33
  Hemoglobin, Day 36, Within, Within | 29 | 32
  Hemoglobin, Day 237, Below, Below: number analyzed (Participants) | 3 | 0
  Hemoglobin, Day 237, Below, Below | 3 |
  Hemoglobin, Day 237, Within, Below: number analyzed (Participants) | 26 | 28
  Hemoglobin, Day 237, Within, Below | 3 | 7
  Hemoglobin, Day 237, Within, Within: number analyzed (Participants) | 26 | 28
  Hemoglobin, Day 237, Within, Within | 23 | 21
  Leukocytes, Day 8, Below, Below: number analyzed (Participants) | 5 | 4
  Leukocytes, Day 8, Below, Below | 2 | 2
  Leukocytes, Day 8, Below, Within: number analyzed (Participants) | 5 | 4
  Leukocytes, Day 8, Below, Within | 3 | 2
  Leukocytes, Day 8, Within, Below: number analyzed (Participants) | 31 | 30
  Leukocytes, Day 8, Within, Below | 2 | 1
  Leukocytes, Day 8, Within, Within: number analyzed (Participants) | 31 | 30
  Leukocytes, Day 8, Within, Within | 28 | 28
  Leukocytes, Day 8, Within, Above: number analyzed (Participants) | 31 | 30
  Leukocytes, Day 8, Within, Above | 1 | 1
  Leukocytes, Day 8, Above, Within: number analyzed (Participants) | 0 | 1
  Leukocytes, Day 8, Above, Within |  | 1
  Leukocytes, Day 36, Below, Below: number analyzed (Participants) | 5 | 4
  Leukocytes, Day 36, Below, Below | 2 | 3
  Leukocytes, Day 36, Below, Within: number analyzed (Participants) | 5 | 4
  Leukocytes, Day 36, Below, Within | 3 | 1
  Leukocytes, Day 36, Within, Below: number analyzed (Participants) | 31 | 29
  Leukocytes, Day 36, Within, Below | 1 | 2
  Leukocytes, Day 36, Within, Within: number analyzed (Participants) | 31 | 29
  Leukocytes, Day 36, Within, Within | 28 | 27
  Leukocytes, Day 36, Within, Above: number analyzed (Participants) | 31 | 29
  Leukocytes, Day 36, Within, Above | 2 | 0
  Leukocytes, Day 36, Above, Above: number analyzed (Participants) | 0 | 1
  Leukocytes, Day 36, Above, Above |  | 1
  Leukocytes, Day 237, Below, Below: number analyzed (Participants) | 4 | 4
  Leukocytes, Day 237, Below, Below | 2 | 1
  Leukocytes, Day 237, Below, Within: number analyzed (Participants) | 4 | 4
  Leukocytes, Day 237, Below, Within | 2 | 3
  Leukocytes, Day 237, Within, Below: number analyzed (Participants) | 25 | 23
  Leukocytes, Day 237, Within, Below | 0 | 1
  Leukocytes, Day 237, Within, Within: number analyzed (Participants) | 25 | 23
  Leukocytes, Day 237, Within, Within | 24 | 21
  Leukocytes, Day 237, Within, Above: number analyzed (Participants) | 25 | 23
  Leukocytes, Day 237, Within, Above | 1 | 1
  Leukocytes, Day 237, Above, Within: number analyzed (Participants) | 0 | 1
  Leukocytes, Day 237, Above, Within |  | 1
  Lymphocytes, Day 8, Unknown, Within: number analyzed (Participants) | 1 | 0
  Lymphocytes, Day 8, Unknown, Within | 1 |
  Lymphocytes, Day 8, Below, Above: number analyzed (Participants) | 0 | 1
  Lymphocytes, Day 8, Below, Above |  | 1
  Lymphocytes, Day 8, Within, Below: number analyzed (Participants) | 35 | 34
  Lymphocytes, Day 8, Within, Below | 1 | 0
  Lymphocytes, Day 8, Within, Within: number analyzed (Participants) | 35 | 34
  Lymphocytes, Day 8, Within, Within | 33 | 34
  Lymphocytes, Day 8, Within, Above: number analyzed (Participants) | 35 | 34
  Lymphocytes, Day 8, Within, Above | 1 | 0
  Lymphocytes, Day 36, Unknown, Within: number analyzed (Participants) | 1 | 0
  Lymphocytes, Day 36, Unknown, Within | 1 |
  Lymphocytes, Day 36, Below, Below: number analyzed (Participants) | 0 | 1
  Lymphocytes, Day 36, Below, Below |  | 1
  Lymphocytes, Day 36, Within, Within: number analyzed (Participants) | 35 | 33
  Lymphocytes, Day 36, Within, Within | 35 | 33
  Lymphocytes, Day 237, Unknown, Within: number analyzed (Participants) | 1 | 0
  Lymphocytes, Day 237, Unknown, Within | 1 |
  Lymphocytes, Day 237, Below, Below: number analyzed (Participants) | 0 | 1
  Lymphocytes, Day 237, Below, Below |  | 1
  Lymphocytes, Day 237, Within, Within: number analyzed (Participants) | 28 | 27
  Lymphocytes, Day 237, Within, Within | 28 | 27
  Monocytes, Day 8, Within, Within: number analyzed (Participants) | 29 | 30
  Monocytes, Day 8, Within, Within | 27 | 25
  Monocytes, Day 8, Within, Above: number analyzed (Participants) | 29 | 30
  Monocytes, Day 8, Within, Above | 2 | 5
  Monocytes, Day 8, Above, Within: number analyzed (Participants) | 7 | 5
  Monocytes, Day 8, Above, Within | 2 | 1
  Monocytes, Day 8, Above, Above: number analyzed (Participants) | 7 | 5
  Monocytes, Day 8, Above, Above | 5 | 4
  Monocytes, Day 36, Within, Within: number analyzed (Participants) | 29 | 29
  Monocytes, Day 36, Within, Within | 25 | 25
  Monocytes, Day 36, Within, Above: number analyzed (Participants) | 29 | 29
  Monocytes, Day 36, Within, Above | 4 | 4
  Monocytes, Day 36, Above, Within: number analyzed (Participants) | 7 | 5
  Monocytes, Day 36, Above, Within | 3 | 1
  Monocytes, Day 36, Above, Above: number analyzed (Participants) | 7 | 5
  Monocytes, Day 36, Above, Above | 4 | 4
  Monocytes, Day 237, Within, Within: number analyzed (Participants) | 24 | 23
  Monocytes, Day 237, Within, Within | 19 | 13
  Monocytes, Day 237, Within, Above: number analyzed (Participants) | 24 | 23
  Monocytes, Day 237, Within, Above | 5 | 10
  Monocytes, Day 237, Above, Within: number analyzed (Participants) | 5 | 5
  Monocytes, Day 237, Above, Within | 0 | 2
  Monocytes, Day 237, Above, Above: number analyzed (Participants) | 5 | 5
  Monocytes, Day 237, Above, Above | 5 | 3
  Neutrophils, Day 8, Below, Within: number analyzed (Participants) | 1 | 0
  Neutrophils, Day 8, Below, Within | 1 |
  Neutrophils, Day 8, Within, Below: number analyzed (Participants) | 35 | 34
  Neutrophils, Day 8, Within, Below | 1 | 4
  Neutrophils, Day 8, Within, Within: number analyzed (Participants) | 35 | 34
  Neutrophils, Day 8, Within, Within | 34 | 29
  Neutrophils, Day 8, Within, Above: number analyzed (Participants) | 35 | 34
  Neutrophils, Day 8, Within, Above | 0 | 1
  Neutrophils, Day 8, Above, Within: number analyzed (Participants) | 0 | 1
  Neutrophils, Day 8, Above, Within |  | 1
  Neutrophils, Day 36, Below, Within: number analyzed (Participants) | 1 | 0
  Neutrophils, Day 36, Below, Within | 1 |
  Neutrophils, Day 36, Within, Below: number analyzed (Participants) | 35 | 33
  Neutrophils, Day 36, Within, Below | 1 | 2
  Neutrophils, Day 36, Within, Within: number analyzed (Participants) | 35 | 33
  Neutrophils, Day 36, Within, Within | 33 | 31
  Neutrophils, Day 36, Within, Above: number analyzed (Participants) | 35 | 33
  Neutrophils, Day 36, Within, Above | 1 | 0
  Neutrophils, Day 36, Above, Within: number analyzed (Participants) | 0 | 1
  Neutrophils, Day 36, Above, Within |  | 1
  Neutrophils, Day 237, Within, Below: number analyzed (Participants) | 29 | 27
  Neutrophils, Day 237, Within, Below | 0 | 1
  Neutrophils, Day 237, Within, Within: number analyzed (Participants) | 29 | 27
  Neutrophils, Day 237, Within, Within | 28 | 25
  Neutrophils, Day 237, Within, Above: number analyzed (Participants) | 29 | 27
  Neutrophils, Day 237, Within, Above | 1 | 1
  Neutrophils, Day 237, Above, Within: number analyzed (Participants) | 0 | 1
  Neutrophils, Day 237, Above, Within |  | 1
  Platelets, Day 8, Below, Below: number analyzed (Participants) | 0 | 1
  Platelets, Day 8, Below, Below |  | 1
  Platelets, Day 8, Within, Within: number analyzed (Participants) | 36 | 34
  Platelets, Day 8, Within, Within | 36 | 34
  Platelets, Day 36, Below, Below: number analyzed (Participants) | 0 | 1
  Platelets, Day 36, Below, Below |  | 1
  Platelets, Day 36, Within, Within: number analyzed (Participants) | 36 | 33
  Platelets, Day 36, Within, Within | 36 | 33
  Platelets, Day 237, Below, Within: number analyzed (Participants) | 0 | 1
  Platelets, Day 237, Below, Within |  | 1
  Platelets, Day 237, Within, Below: number analyzed (Participants) | 29 | 27
  Platelets, Day 237, Within, Below | 0 | 1
  Platelets, Day 237, Within, Within: number analyzed (Participants) | 29 | 27
  Platelets, Day 237, Within, Within | 29 | 25
  Platelets, Day 237, Within, Above: number analyzed (Participants) | 29 | 27
  Platelets, Day 237, Within, Above | 0 | 1

16. Secondary Outcome: Anti-S. Sonnei Lipopolysaccharide (LPS) Immunoglobulin G (IgG) Antibody Concentrations at Pre-vaccination and After the First and Second Vaccination
Description: Anti-S. sonnei LPS IgG antibody concentrations are presented as geometric mean concentrations (GMCs), determined by Enzyme-linked immunosorbent assay (ELISA) and expressed in ELISA units per milliliter (EU/mL). Note: regarding the "28 days after second vaccination" protocol timing, sample collection could have been performed either at Day 56 or at Day 57. For all the subjects, samples were collected at Day 56, and therefore, results are presented for "Day 56 (27 days after the second vaccination)" timing.
Time Frame: At Day 1 (pre-vaccination), at Day 8 (7 days after the first vaccination), at Day 29 (28 days after the first vaccination), at Day 36 (7 days after the second vaccination) and at Day 56 (27 days after the second vaccination)
Population: The analysis is performed on the Per protocol Set for immunogenicity, which includes all subjects who correctly received the study vaccine or placebo, have no protocol deviations leading to exclusion and provide post-vaccination immunogenicity data at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 34 | 31
EU/mL
  Day 1 | 99.32 [62.39 to 158.11] | 124.07 [77.30 to 199.13]
  Day 8 | 229.18 [135.69 to 387.09] | 128.24 [81.43 to 201.96]
  Day 29 | 523.21 [304.08 to 900.24] | 124.48 [76.16 to 203.46]
  Day 36 | 577.86 [345.36 to 966.90] | 123.57 [77.31 to 197.50]
  Day 56 | 548.75 [325.13 to 926.18] | 134.24 [85.12 to 211.70]

17. Secondary Outcome: Anti-S. Sonnei LPS IgG Antibody Concentrations at Pre-challenge and After Challenge
Description: Anti-S. sonnei LPS IgG antibody concentrations are presented as GMCs, as determined by ELISA and expressed in EU/mL. Note: regarding the "28 days after second vaccination" protocol timing, sample collection could have been performed either at Day 56 or at Day 57. For all the subjects, samples were collected at Day 56, and therefore, results are presented for "Day 56 (27 days after the second vaccination)" timing.
Time Frame: At Day 56 (pre-challenge), at Day 64 (7 days after challenge) and at Day 85 (28 days after challenge)
Population: The analysis is performed on the Per protocol Set for immunogenicity, which includes all subjects who correctly received the study vaccine or placebo and challenge agent, have no protocol deviations leading to exclusion and provide post-vaccination immunogenicity data at the specified time points.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 30 | 26
EU/mL
  Day 56 | 529.4 [296.83 to 944.20] | 150.59 [90.55 to 250.42]
  Day 64 | 537.92 [295.66 to 978.71] | 216.11 [132.83 to 351.61]
  Day 85 | 1039.07 [601.00 to 1796.46] | 810.97 [419.53 to 1567.65]

18. Secondary Outcome: Number of Subjects Achieving a Post-vaccination Anti-S. Sonnei LPS Concentration ≥ 268 EU/mL
Description: This antibody response cut-off was based on the results of the previous Phase I studies and estimated results of the median antibody titer after natural infection by S. sonnei. The threshold 121 EU/mL planned per protocol has been recalibrated to 268 EU/mL following an investigation of reliability of the ELISA assay. Note: regarding the "28 days after second vaccination" protocol timing, sample collection could have been performed either at Day 56 or at Day 57. For all the subjects, samples were collected at Day 56, and therefore, results are presented for "Day 56 (27 days after the second vaccination)" timing.
Time Frame: At Day 29 (28 days after the first vaccination) and at Day 56 (27 days after the second vaccination)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 34 | 31
Participants
  Day 29 | 24 | 7
  Day 56 | 24 | 7

19. Secondary Outcome: Number of Seroresponders for Anti-S. Sonnei LPS
Description: Seroresponse definition as reported in the protocol was assay specific and specifically related to assay, as run in Marburg Lab for the previous GVGH Shigella studies. This assay was further characterized and optimized before being used in GVGH for the current Phase 2b study. Since the assay used in current study is not comparable with the assay used in previous GVGH studies, the seroresponse definition is no longer appropriate (as it is valid only for Marburg assay). With the acknowledgment that seroresponse results are no longer meaningful, the study team choose to report the results for transparency. Note: regarding the "28 days after second vaccination" protocol timing, sample collection could have been performed either at Day 56 or at Day 57. For all the subjects, samples were collected at Day 56, and therefore, results are presented for "Day 56 (27 days after the second vaccination" timing.
Time Frame: At Day 29 (28 days after the first vaccination) and at Day 56 (27 days after the second vaccination)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | S. Sonnei Group | Placebo Group
Number analyzed (Participants) | 34 | 31
Participants
  Day 29 | 32 | 0
  Day 56 | 31 | 0

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected within the 7-day post-vaccination period or 8-day post-challenge period. Unsolicited AEs were collected within the 28-day post-vaccination or post-challenge period. SAEs were collected from Day 1 up to study end at Day 237.
Arm/Group | S. Sonnei Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/35
Other Adverse Events (participants affected / at risk) | 34/36 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S. Sonnei Group (N=36) | Placebo Group (N=35)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | S. Sonnei Group (N=36) | Placebo Group (N=35)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 18 (23) | 15 (18)
Aphthous ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 22 (23) | 22 (22)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 13 (13) | 16 (16)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (11) | 10 (11)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (7) | 4 (4)
Chills (General disorders) | 12 (15) | 5 (7)
Fatigue (General disorders) | 13 (18) | 12 (15)
Induration (General disorders) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 31 (54) | 13 (17)
Malaise (General disorders) | 19 (29) | 16 (24)
Pyrexia (General disorders) | 4 (4) | 5 (5)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 1 (1)
Anal injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 2 (3) | 5 (7)
Decreased appetite (Metabolism and nutrition disorders) | 14 (14) | 13 (13)
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 (24) | 10 (14)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (35) | 16 (28)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 22 (31) | 22 (29)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 3 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-07-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT03527173/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-03): https://cdn.clinicaltrials.gov/large-docs/73/NCT03527173/SAP_001.pdf